CLINICAL TRIAL: NCT03994744
Title: A Phase II Open-label, Single-arm Study Assessing the Efficacy and Safety of Combination Therapy of Sintilimab and Metformin With Relapsed PD-L1 Positive Small Cell Lung Cancer
Brief Title: Assessing Safety and Efficacy of Sintilimab and Metformin Combination Therapy in SCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hunan Cancer Hospital (Other)
Collaborators: Xiangya Hospital of Central South University (Other); Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Principal Investigator, Lin Wu, Chief physician, director of department, Hunan Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HNCH-SCLC-2019260
Record Dates: First submitted 2019-06-19; First posted 2019-06-21 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Small-cell Lung Cancer; Small Cell Lung Carcinoma; Small Cell Lung Cancer Recurrent; Small Cell Lung Cancer Extensive Stage
Keywords: immunotherapy; metformin; PD-L1; PD-1 checkpoint inhibitor
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Immune Checkpoint Inhibitors; sintilimab; Metformin

STUDY DESIGN:
Intervention Model Description: Patients fulfilling Eligibility Criteria will be included in our study. Participants will be given intravenous administration of Sintilimab (1200mg/3w).
  Metformin treatment will be given (day20) 1 week before the second administration of Sintilimab at a dose of 2000 mg daily (1000mg BID).
  Treatments will be administrated for one year or until disease progression, death, or unacceptable toxicity.
  Regular follow-up and safety assessment: Patients were assessed for drug safety and treatment efficacy every 2 cycles (6 weeks) in the first 3 months after enrollment, and then evaluated every 4 cycles (12 weeks). Assessment of tumor response, adverse events. Follow-up until disease progression and patient death.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sintilimab and Metformin (Experimental): Participants will be given intravenous administration of Sintilimab (1200mg/3w) Metformin treatment will be given (day20) 1 week before the second administration of Sintilimab a a dose of 2000 mg daily (1000mg BID).
  The duration of treatment will be up to one year, or till the disease progression, death, or unacceptable toxicity show up.
  Interventions: Drug: PD-1 inhibitor; Drug: Metformin

INTERVENTIONS:
Drug: PD-1 inhibitor — Intravenous administration of Sintilimab (1200mg/3weeks)
  Other Names: Sintilimab; IBI380
Drug: Metformin — Metformin treatment will be given (day20) 1 week before the second administration of Sintilimab at a dose of 2000 mg daily (1000mg BID).
  To reduce GI toxicity, participants start Metformin at 1000 mg daily (500mg am, 500 mg pm) for 1 week.

SUMMARY:
In this Single arm study, histologically or cytologically confirmed ED-stage small cell lung cancer (SCLC) patients resistant to or relapsed after standard chemotherapy will be enrolled to investigate the Efficacy and Safety of a Combination of Sintilimab and Metformin.

Primary outcome:

Objective response rate (ORR), Safety of the combination therapy

Secondary outcome:

Overall survival (OS), Progression-free survival (PFS), Duration of response(DOR),

DETAILED DESCRIPTION:
Exploratory Endpoints:

The association between the efficacy of the combination treatment and changes in CTC counts after administration of the treatment.

Evaluating the correlation between programmed death ligand 1 (PD-L1) expression derived from circulating tumor cells (CTC) and tumor tissue cells, and the predictive role of CTC PD-L1 expression in ED-SCLC.

The compositional changes in the gut microbiota after administration of the treatment and its association with the efficacy of the combination treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient, age≥18 and≤65;
2. Eastern Cooperative Oncology Group (ECOG) performance status ≤2;
3. The life expectancy of greater than 12 weeks;
4. Participants must have histologically or cytologically confirmed metastatic or extended disease of SCLC (ED-SCLC).
5. According to RECIST1.1, participants must have been confirmed Disease progression (within 6 months, confirmed by imaging test)after platinum-based doublet chemotherapy OR after (PFS>6 months, ) platinum-based doublet chemotherapy and refused to continue chemotherapy, OR after second-line or more lines of systemic chemotherapy limited disease SCLC (LD-SCLC) patients with disease progression after Synchronous chemoradiotherapy, must receive firstline systematic platinum-based doublet chemotherapy and refused to receive chemotherapy again.
6. Evaluable or measurable lesion is required, defined as at least one lesion (not brain metastasis) that can be accurately measured based on RECIST 1.1;
7. Participant need to provided tumor tissue (from an archival tumor sample obtained within 1 year or from a new biopsy sample) for PD-L1 immunohistochemical (IHC) assay, and PD-L1expression in more than 1% cells is required;
8. Participant is able to the ability to swallow oral medications
9. Participants have to meet the following criteria to ensure function of vital organs:

   Absolute neutrophil count (ANC) ≥1.5×109/L or White blood cell count >3.5×109/L;Platelets >80×109/L; Hemoglobin (HGB)≥90 g/L;Serum total bilirubin ≤ 1.5 x upper limit of normal (ULN); AST(SGOT)/ALT(SGPT) ≤2.5 ×ULN; ALB≥2.8g/dL;Serum creatinine ≤ 1.5 x institutional ULN OR creatinine clearance ≥40 mL/min using the Cockcroft-Gault equation
10. Participants must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) through the treatment, and for at least 180 days after the last dose of study treatment; Participants must have the ability to understand and be willing to sign a written informed consent document.

Exclusion Criteria:

1. Participants who were diagnosed as mixed pathological type of small cell lung cancer
2. Participants who had long-term use of metformin (>2 weeks) 6 months prior to study entry, or diagnosed with type-2 diabetes,
3. Participants received treatment with anti-PD1, -PDL1, -CTLA4, -CD137 inhibitors before, or any therapy specifically targeting T-cell co-stimulation or checkpoint pathways.
4. Participants received cellular immunotherapy before
5. Participants with Uncontrolled intercurrent illness including, but not limited to:

   Ongoing or active infection; Known history of Human Immunodeficiency Virus (HIV) infection Acute or chronic active hepatitis B (HBV DNA >1*10^3 copies/ml or >200 IU/mL) or, acute or chronic active hepatitis C (with a positive Hepatitis C antibody test result) Active tuberculosis Congestive heart failure (Class III-IV, according to New York Heart Association classification), or and clinically significant Cardiac arrhythmia if poorly controlled; Uncontrolled arterial hypertension (systolic blood pressure ≥160mmHg or diastolic blood pressure ≥100mmHg) Any arterial thrombosis, embolism, ischemia, myocardial infarction, unstable angina, or cerebrovascular accident within 6 months prior to enrollment,
6. Participants with symptomatic Central nervous metastasis or meningeal carcinomatosis are excluded; Participants with asymptomatic brain metastases or with brain metastases that have been treated and stable in a subsequent scan are allowed to include if there is measurable lesion outside the Central nervous system and no history of intracranial hemorrhage, and not midbrain, pons, cerebellum, medulla or spinal cord metastasis, and do not need glucocorticoid therapy.
7. Participants receiving glucocorticoid (>30 mg prednisone equivalent a day) or any Immunosuppressive drug within 14 days prior to study recruitment; Participants receiving inhaled or Topical corticosteroids, adrenal corticosteroid replacement therapy (>10 mg prednisone equivalent a day) are allowed if they have no active autoimmune disease
8. Participants with a known additional malignancy (Except for Non-melanoma skin cancer and the following in situ carcinoma: in situ bladder carcinoma, in situ gastric carcinoma, in situ colonic carcinoma, in situ endometrial carcinoma, in situ cervical carcinoma /dysplasia, in situ melanoma carcinoma and in situ breast Carcinoma) unless they Maintained Complete Remission for at least 5 years and do not need corresponding treatment during the study
9. Participants who have not recovered (i.e., ≤ Grade 1 according to NCI CTCAE V4or at baseline) from adverse effects due to a previously administered agent.
10. Participants who have uncontrollable effusion, such as pleural and ascites that cannot be controlled by drainage or other treatment
11. Patients who have active autoimmune diseases; excluding patients whose active autoimmune disease is caused by Vitiligo or asthma that is completely relieved in childhood and Patients with hypothyroidism requiring only hormone replacement therapy
12. Patients with known Allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation
13. Patients who are pregnant or breastfeeding,
14. Patients who are allergic to monoclonal antibody drugs
15. Patients who have contraindications to metformin including severe allergic reactions and intolerance
16. Patients who are not eligible for this study, as Assessed by Investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2019-08-20 (Actual); Primary Completion 2021-08-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate of Sintilimab and Metformin(ORR) | 1 year
  Assessing the response of treatment of each patient using RECIST 1.1 criteria, the investigators calculate the percentage of patients meet partial response (30% decrease in diameter) and complete response in the arm.
Safety of the combination therapy of Sintilimab and Metformin: CTCAE4.03 grading | 2 year
  Incidence and severity of (serious) adverse events in each individual according to the CTCAE4.03 grading.

SECONDARY OUTCOMES:
Median overall survival (OS) time of Sintilimab and Metformin | 2 years
  Use K-M to estimate the median OS of single arm.
Median progression free survival(PFS) of Sintilimab and Metformin | 1 year
  Use K-M to estimate the median PFS of single arm.
Median duration of response (DoR) of Sintilimab and Metformin | 1 year
  Use K-M to estimate the median DoR of single arm.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Wu, Principal Investigator — Hunan Cancer Hospital
Locations (1):
- Hunan Cancer hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: please contact the principal investigator of this study or correspondence author of published wotk.

REFERENCES:
- [Derived] Aden D, Sureka N, Zaheer S, Chaurasia JK, Zaheer S. Metabolic Reprogramming in Cancer: Implications for Immunosuppressive Microenvironment. Immunology. 2025 Jan;174(1):30-72. doi: 10.1111/imm.13871. Epub 2024 Oct 27. PMID 39462179